CLINICAL TRIAL: NCT02319356
Title: Does Dietary Nitrate Supplementation Improve Aerobic Performance in Colorectal Cancer? A Pilot Study
Brief Title: Does Dietary Nitrate Supplementation Improve Aerobic Performance
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Vanessa Brown, Responsible research fellow, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 163841
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Beetroot juice (BRJ) (Active Comparator): beetroot juice
  Interventions: Dietary Supplement: Beetroot juice
- Placebo (PL) (Placebo Comparator): placebo juice
  Interventions: Dietary Supplement: Placebo beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — (BRJ, containing NO3-, 6.2 mmol/day, administered as 500ml Beet it Sport Shots, James White drinks, Ipswich uk)
  Other Names: Beet it Sport Shots
  Arms: Beetroot juice (BRJ)
Dietary Supplement: Placebo beetroot juice — (PL, NO3-depleted beetroot juice, administered as 500ml Placebo Beet it Sport Shots, James White drinks, Ipswich uk)
  Other Names: Nitrate deplete Beet it Sport Shots
  Arms: Placebo (PL)

SUMMARY:
The purpose of this study is to determine whether dietary nitrate supplementation improves performance in cardiopulmonary exercise testing (CPET).

DETAILED DESCRIPTION:
Dietary nitrate supplementation has been shown to enhance exercise tolerance and performance in professional athletes and physically active males.

Cardiopulmonary exercise testing (CPET) is an established, non invasive and safe method of assessing patients' cardiopulmonary reserve prior to surgery. It has been shown to predict complications and length of stay in patients undergoing major elective surgery.

The anaerobic threshold (AT), the oxygen uptake at which anaerobic ATP synthesis supplements aerobic ATP synthesis and the maximal oxygen uptake (VO2max) the point where the oxygen uptake plateaus despite an increase in work rate; both calculated during CPET; have both been shown to predict short and long term outcomes after surgery and postoperative complications.

We aim to study the effect of dietary nitrate supplementation on CPET results in patients awaiting surgery for colorectal cancer.

Our primary outcome will be the change in the AT and VO2Max after beetroot juice supplementation.

Methods: Patients will undergo an initial CPET and will then be randomized to receive either beetroot juice (BRJ, containing NO3-, 6.2 mmol/day, administered as 500ml Beet it Sport Shots, James White drinks, Ipswich uk) or 'placebo' (PL, NO3-depleted beetroot juice) for 7 days. A second CPET will then be performed.

This pilot study will be used to calculate the mean AT and VO2Max and associated standard deviations for our population and the approximate effect of BRJ on them.

ELIGIBILITY:
Inclusion Criteria:

* Elective Colonic or rectal resection.

Exclusion Criteria:

* Contraindication to cardiopulmonary exercise testing: unstable cardiac disease, lower limb dysfunction, inability to perform CPET
* Inability to give informed consent
* Emergency surgery
* During CPET: Ischemic ECG or inability to reach AT
* Allergy to Beetroot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
anaerobic threshold (AT) | 1 year
  The change in the anaerobic threshold (AT) after beetroot juice supplementation.
maximal oxygen uptake (VO2Max) | 1 year
  The change in the maximal oxygen uptake (VO2Max) after beetroot juice supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Brown, MBBS, MRCS, Principal Investigator — Royal Surrey County Hospital Guildford

REFERENCES:
- [Background] Jones AM. Dietary nitrate supplementation and exercise performance. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S35-45. doi: 10.1007/s40279-014-0149-y. PMID 24791915
- [Background] Snowden CP, Prentis JM, Anderson HL, Roberts DR, Randles D, Renton M, Manas DM. Submaximal cardiopulmonary exercise testing predicts complications and hospital length of stay in patients undergoing major elective surgery. Ann Surg. 2010 Mar;251(3):535-41. doi: 10.1097/SLA.0b013e3181cf811d. PMID 20134313
- [Background] Colson M, Baglin J, Bolsin S, Grocott MP. Cardiopulmonary exercise testing predicts 5 yr survival after major surgery. Br J Anaesth. 2012 Nov;109(5):735-41. doi: 10.1093/bja/aes263. Epub 2012 Aug 21. PMID 22910977